CLINICAL TRIAL: NCT03704142
Title: Personal Amplification Devices in Noise and Speech Maskers
Brief Title: Comparison of PSAPs in Different Maskers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Karen Helfer, Principal Investigator, University of Massachusetts, Amherst
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMassAmherst
Record Dates: First submitted 2018-09-06; First posted 2018-10-12 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-02

CONDITIONS: Auditory Perception

STUDY DESIGN:
Intervention Model Description: Each participant will be tested with one of the models of devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tweak Focus (Experimental): Speech understanding and listening effort will be assessed using the Tweak Focus personal sound amplifiers.
  Interventions: Device: Tweak Focus
- IQ Earbuds (Experimental): Speech understanding and listening effort will be assessed using the IQEarbuds personal sound amplifiers.
  Interventions: Device: IQ Earbuds
- Sound World Solutions CS50+ (Experimental): Speech understanding and listening effort will be assessed using the Sound World Solutions CS50+ personal sound amplifiers.
  Interventions: Device: Sound World Solutions CS50+
- Bose Hearphones (Experimental): Speech understanding and listening effort will be assessed using the Sound World Solutions CS50+ personal sound amplifiers.
  Interventions: Device: Bose Hearphones

INTERVENTIONS:
Device: Sound World Solutions CS50+ — Participants will be tested using the Sound World Solutions CS 50+ hearing devices.
  Arms: Sound World Solutions CS50+
Device: Tweak Focus — Participants will be tested using the Tweak Focus hearing devices.
  Arms: Tweak Focus
Device: IQ Earbuds — Participants will be tested using the IQ Earbuds hearing devices.
  Arms: IQ Earbuds
Device: Bose Hearphones — Participants will be tested using the Bose Hearphones hearing devices.
  Arms: Bose Hearphones

SUMMARY:
This study will measure the performance of three personal amplification devices when used by middle-aged adults. Speech understanding will be assessed with two different types of background noises at three different input levels.

DETAILED DESCRIPTION:
Speech understanding will be measured both unaided and aided with three different models of Personal Amplification devices (PSAPs). Sentences will be played to the participant from a loudspeaker located in front. Different types of background sounds (noise and other sentences) will be played from loudspeakers located to the right and left of the participant. Participants will be instructed to repeat back the sentence coming from the front. They also will rate subjective effort at the end of each block of trials.

ELIGIBILITY:
Inclusion Criteria:

* mild high-frequency hearing loss (pure-tone thresholds of 25 decibels hearing loss - 45 decibels hearing loss between 2000 Hz and 6000 Hz)

Exclusion Criteria:

* history of prior hearing aid use
* history of neurologic or otologic disorders
* score of < 26 on Montreal Cognitive Assessment (cognitive screening tool)

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tweak Focus | IQ Earbuds | Sound World Solutions CS50+ | Bose Hearphones
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tweak Focus | IQ Earbuds | Sound World Solutions CS50+ | Bose Hearphones | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (4.01) | 58.4 (5.46) | 59.6 (4.06) | 57 (4.11) | 58.4 (4.38)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Reported gender: Female | 5 | 9 | 7 | 6 | 27
  Reported gender: Male | 5 | 0 | 3 | 4 | 12
  Reported gender: Other/not reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 10 | 40
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40
Hearing loss (better-ear high-frequency pure tone average) [Mean (Standard Deviation); unit: Decibels Hearing Loss] — Level of hearing loss, determined by puretone audiometry; average hearing loss in better ear for frequencies 2000-6000 Herz
  Decibels Hearing Loss | 22 (13.41) | 23.5 (9.57) | 23.5 (11.13) | 20.13 (13.83) | 22.28 (11.72)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of How Four Models of Personal Listening Devices Improve Word Understanding in Noise
Description: Improvement in performance on speech perception task using the Nuheara IQ Buds, Tweak Focus, Bose Hearphones, or the Sound World Solutions CS 50+ personal listening devices, measured by percentage of words accurately recalled in noise with device minus percentage recalled without device. Positive values indicate improvement in performance.
Time Frame: One 2-hour lab session
Measure: Mean (Standard Deviation); unit: Percent of words recalled
Groups:
- Tweak Focus: Group of participants assigned to use the Tweak Focus hearing device
- CS50+: Group of participants who were assigned the Sound World Solutions CS50+ listening device
- IQ Buds: Group of participants who were assigned the Nuheara IQ Buds listening device
- Bose: Group of participants who were assigned the Bose Hearphones listening device
Arm/Group | Tweak Focus | CS50+ | IQ Buds | Bose
Number analyzed (Participants) | 10 | 10 | 10 | 10
Percent of words recalled | 1.65 (6.40) | 0.85 (7.01) | 7.35 (6.03) | 10.24 (8.23)

2. Secondary Outcome: Difference in Self-rated Listening Effort
Description: Effect of listening devices on subjective listening effort, measured by rating on ten-point scale (10 = greatest amount of effort) after task performed with device minus rating after task performed without device. Lower scores indicate less listening effort; negative values indicate reduction in effort with device.
Time Frame: One 2-hour session
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tweak Focus | CS50+ | IQ Buds | Bose
Number analyzed (Participants) | 10 | 10 | 10 | 10
Units on a scale | -1.4 (1.26) | -1.4 (1.84) | -0.9 (1.29) | -1.8 (1.81)

ADVERSE EVENTS:
Time Frame: Lab visit (1-3 hours)
Arm/Group | Tweak Focus | IQ Earbuds | Sound World Solutions CS50+ | Bose Hearphones
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT03704142/Prot_SAP_ICF_000.pdf